CLINICAL TRIAL: NCT00148525
Title: Trial of 2 TeleComputer Diet Change Maintenance Programs
Brief Title: The Study of Automated Telephone Programs for the Maintenance of Dietary Change
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert H. Friedman (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Robert H. Friedman, Professor of Medicine, Boston Medical Center
Organization: Boston Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CA105832-02 (NIH); National Cancer Institute
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2011-06

CONDITIONS: Cancer
Keywords: automated telephony, cancer prevention, healthy diet
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- social cognitive theory (Experimental): This arm received an diet intervention designed to maintain changes in fruit and vegetable consumption. The intervention components were based on social cognitive theory and delivered by an automated telephone system.
  Interventions: Behavioral: Social Cognitive Theory
- Goal Systems Theory (Experimental): This arm received an diet intervention designed to maintain changes in fruit and vegetable consumption. The intervention components were based on goal systems theory.
  Interventions: Behavioral: goal system theory
- Comparison group (No Intervention): comparison group

INTERVENTIONS:
Behavioral: Social Cognitive Theory — 6 mo dietary intervention. This arm received an diet intervention designed to maintain changes in fruit and vegetable consumption. The intervention components were based on social cognitive theory.
  Other Names: Social cognitive theory (SCT)
  Arms: social cognitive theory
Behavioral: goal system theory — This arm received a 6 mo diet intervention designed to maintain changes in fruit and vegetable consumption. The intervention components were based on goal systems theory and delivered by an automated telephone system.
  Other Names: Goal systems theory (GST)
  Arms: Goal Systems Theory

SUMMARY:
The purpose of this study is to test two different approaches to helping individuals who have recently starting eating a healthful diet maintain those healthy changes. This study will deliver a health program using an automated telephone system. The programs will be designed to help individuals maintain a healthy diet change for a lifetime.

DETAILED DESCRIPTION:
RCT is completed. However, the eligibility was 18 y/o or greater and living in Greater Boston area. The participants used an evidenced based dietary intervention for 3 months and then were randomized to 1 of 3 arms. Those in the experimental arm received a 6 mo intervention based on social cognitive theory or goal systems theory. The intervention was designed to help the participants maintain previously achieved changes in the their diet, e.g., fruits and vegetables. The outcome measures are fruit and vegetable consumption as measured by servings on multiple dietary measures as well as a 24 hr dietary recall.

ELIGIBILITY:
Inclusion Criteria:

* Consume fewer than 5 fruits and vegetables per day.
* Understand conversational English
* Have the ability to use a telephone without assistance

Exclusion Criteria:

* Under 18 years of age
* Diagnosis of a health condition for which dietary recommendations in the would be contraindicated,
* Have cognitive impairment
* Have a terminal illness, recent myocardial infarction, current or former diagnosis of an eating disorder, pregnancy
* Consume > 5 servings of fruit and vegetable per day, or
* Plan to move away from the Boston area in less than 30 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2006-07; Primary Completion 2010-08 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The study hypothesis is that the goal systems intervention will out perform the social cognitive intervention and that both of these interventions will outperform the control group for fruit and vegetable consumption. | July 2006-July 2009

SECONDARY OUTCOMES:
Intervention effects will be mediated by behavioral factors predicted by Social Cognitive Theory and Goal Systems Theory. | July 2006-July 2009

CONTACTS AND LOCATIONS:
Overall Officials: Robert Friedman, MD, Principal Investigator — Boston University
Locations (1):
- Boston medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wright JA, Quintiliani LM, Turner-McGrievy GM, Migneault JP, Heeren T, Friedman RH. Comparison of two theory-based, fully automated telephone interventions designed to maintain dietary change in healthy adults: study protocol of a three-arm randomized controlled trial. JMIR Res Protoc. 2014 Nov 10;3(4):e62. doi: 10.2196/resprot.3367. PMID 25387065